CLINICAL TRIAL: NCT03544619
Title: Reliability and Cross-cultural Adaptation of the Turkish Version of the Neuropathic Pain Symptom Inventory
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Erenköy Physical Therapy and Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, AYLİN SARI, Medical doctor, specialist on physical therapy and rehabilitation, Erenköy Physical Therapy and Rehabilitation Hospital
Other Study IDs: AYLIN2
Record Dates: First submitted 2018-05-21; First posted 2018-06-04 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neuropathic Pain Symptom Inventory — Investigators will use the Neuropathic Pain Symptom Inventory for assessing neuropathic symptoms

SUMMARY:
In this study, investigators want to perform the reliability and cross-cultural Adaptation of the Turkish Version of the Neuropathic Pain Symptom Inventory

DETAILED DESCRIPTION:
The purpose of the study is to determine the Turkish version, the reliability and cross-cultural Adaptation of the Turkish Version of the Neuropathic Pain Symptom Inventory. 120 patients with neuropathic pain will be included in the study. Test-retest and internal consistency analysis were conducted to determine the reliability of the questionnaire. Test-retest results evaluated using the Intraclass Correlation Coefficient method.

ELIGIBILITY:
Inclusion Criteria:

* Age upper 18
* Complaints of neuropathic pain for at least 3 months

Exclusion Criteria:

* Presence of psychiatric illness
* Cancer pain, unsuccessful lumbar surgeon syndrome etc. mix type pain presence
* Presence of complex regional pain syndrome
* Cognitive impairment (mini-mental test score <24)
* Native language is not Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have neuropathic symptoms
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-06-10 (Actual); Primary Completion 2020-12-25 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Reliability and adaptation | 7 weeks
  Investigators will use linguistic validaiton guideline of Mapi research.
DN4 | 5 minutes
  DN4 has become one of the principal condition-specific outcome measures of neuropathic pain.Investigators will use it for comparing results of NPSI.

CONTACTS AND LOCATIONS:
Overall Officials: unsal sarı, Study Chair — ERENKOY PHYSICAL THERAPY AND REHABILITATION HOSPITAL
Locations (1):
- Erenkoy Physical Treatment Nad Rehabilitation Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No